CLINICAL TRIAL: NCT02643407
Title: Nedaplatin/Docetaxel Versus Cisplatin/Docetaxel in Treatment of Advanced/Relapsed Squamous Cell Lung Cancer :A Randomized, Open, Parallel, Multicentre, Phase Ⅲ Study
Brief Title: Nedaplatin/Docetaxel Versus Cisplatin/Docetaxel in Treatment of Advanced/Relapsed Squamous Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, MD, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1501
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: squamous cell carcinoma; nedaplatin; cisplatin; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — Docetaxel; nedaplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel plus Nedaplatin (Experimental): docetaxel 60mg/m2 and nedaplatin 80mg/m2, d1 every 3 weeks
  Interventions: Drug: Docetaxel; Drug: Nedaplatin
- Docetaxel plus Cisplatin (Active Comparator): docetaxel 60mg/m2 and cisplatin 75mg/m2, d1 every 3 weeks
  Interventions: Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — 60mg/m2
Drug: Nedaplatin — 80mg/m2
  Arms: Docetaxel plus Nedaplatin
Drug: Cisplatin — 75mg/m2
  Arms: Docetaxel plus Cisplatin

SUMMARY:
To compare the efficacy and safety of docetaxel plus nedaplatin with docetaxel plus cisplatin in managment of advanced/relapsed squamous cell lung cancer.

DETAILED DESCRIPTION:
This study is prospective to evaluate whether the efficacy and safety of docetaxel plus nedaplatin is non-inferior to docetaxel plus cisplatin in managment of advanced/relapsed squamous cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were required to be between 18 to 75 years, with histologically or cytologically proven squamous cell carcinoma of the lung, stage ⅢB (unfit for definitive radiotherapy), stage Ⅳ or relapsing;
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of zero or one;
3. life expectancy > 3 months;
4. No previous history of malignancy (except adequately treated carcinoma-in-situ of the cervix or basal cell carcinoma of the skin or superficial bladder cancer [Ta, Tis & T1]); previously untreated with chemotherapy (eg. gemcitabine, platinum, paclitaxel); no previously systemic therapy on locally advanced and metastatic disease; patients were eligible for participation in the study if they had recurrence or metastasis and became locally advanced or metastatic lung cancer after 12 months treatment with gemcitabine, platinum or paclitaxel regimen in adjuvant or neoadjuvant chemotherapy;
5. Adequate organ function was required, as evidenced by absolute neutrophil count ≥ 1.5 x 109 /L, platelet count ≥ 100 x109/L, hemoglobin ≥ 90 g/L (9 g/dL);
6. hepatic enzyme levels ≤ 2.5 x the upper limit of the normal range (ULN), alkaline phosphatase levels ≤ 5.0 x the ULN, total bilirubin levels ≤ 1.5 x the ULN, and serum creatinine levels ≤1.5 mg/dL (or creatinine clearance ≥50 mL/min);
7. Previous radiotherapy was allowed if it involved <25% of bone marrow and was completed 4 weeks before study entry; Patients must be recovered from acute toxicity before the clinical trials;
8. Pregnancy test: negative (female only); Women with fertility need pregnancy test (serum or urine) in 7 days before entering the group and the results were negative. Male or female patients with reproduction potential had to use an approved contraceptive method during and for 8 weeks after the end of study treatment.
9. Patients are judged by researcher to be the compliance of research requirements and follow-up.
10. All the patients provided their written informed consent before enrollment.
11. The standard first-line platinum-based regimens according to the clinical practice, and the efficacy was evaluated every two cycles.

Exclusion Criteria:

1. EGFR positive or ALK positive (patients, the status of EGFR and ALK were unknown due to the detection, were included);
2. Participation in any clinical research in 4 weeks before the first dosage, except non interventional epidemiological investigation;
3. Patients with the complications in high risk;
4. Primary brain tumors or central nervous system (CNS) metastatic carcinoma. The patients who are suspected the CNS metastatic carcinoma should be scanned in 28 days before entering the group. Other malignant disease five years ago (except cone-biopsied carcinoma-in-situ of the cervix or adequately treated basal or squamous cell carcinoma of the skin)
5. Third-space fluid collection that has the clinical significance, such as ascites or pleural effusion, cannot control through the drainage or other method;
6. Serious mental retardation or cognitive impairment, psychotic illness, poor compliance, cannot meet and narrate therapy responders;
7. No eliminated acute or chronic infection, or other serious concomitant diseases;
8. Serious or uncontrolled concomitant disorders (active infection, ischemic heart diseases, arrhythmia, liver dysfunction, or peripheral nerve disorder);
9. Patients with bleeding tendency or organ transplant;
10. Alcohol or drug dependent patients; patients with the chronic administration of adrenal cortical hormone or immunosuppressive; patients with AIDS or other infectious diseases;
11. Active hepatitis, liver metastasis is over 3/4 of the whole liver;
12. A history of drug allergy;
13. The female patients in the reproductive years are unwilling contraception;
14. Accept other anti-tumor therapy at the same time;
15. The researchers believe that the patients are not able to complete the entire clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Li T, Kung HJ, Mack PC, Gandara DR. Genotyping and genomic profiling of non-small-cell lung cancer: implications for current and future therapies. J Clin Oncol. 2013 Mar 10;31(8):1039-49. doi: 10.1200/JCO.2012.45.3753. Epub 2013 Feb 11. PMID 23401433
- [Background] Mitsudomi T, Yatabe Y. Mutations of the epidermal growth factor receptor gene and related genes as determinants of epidermal growth factor receptor tyrosine kinase inhibitors sensitivity in lung cancer. Cancer Sci. 2007 Dec;98(12):1817-24. doi: 10.1111/j.1349-7006.2007.00607.x. Epub 2007 Sep 20. PMID 17888036
- [Background] Soda M, Choi YL, Enomoto M, Takada S, Yamashita Y, Ishikawa S, Fujiwara S, Watanabe H, Kurashina K, Hatanaka H, Bando M, Ohno S, Ishikawa Y, Aburatani H, Niki T, Sohara Y, Sugiyama Y, Mano H. Identification of the transforming EML4-ALK fusion gene in non-small-cell lung cancer. Nature. 2007 Aug 2;448(7153):561-6. doi: 10.1038/nature05945. Epub 2007 Jul 11. PMID 17625570
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Hoang T, Dahlberg SE, Schiller JH, Johnson DH. Does histology predict survival of advanced non-small cell lung cancer patients treated with platin-based chemotherapy? An analysis of the Eastern Cooperative Oncology Group Study E1594. Lung Cancer. 2013 Jul;81(1):47-52. doi: 10.1016/j.lungcan.2013.03.018. Epub 2013 Apr 21. PMID 23611404
- [Background] Fossella F, Pereira JR, von Pawel J, Pluzanska A, Gorbounova V, Kaukel E, Mattson KV, Ramlau R, Szczesna A, Fidias P, Millward M, Belani CP. Randomized, multinational, phase III study of docetaxel plus platinum combinations versus vinorelbine plus cisplatin for advanced non-small-cell lung cancer: the TAX 326 study group. J Clin Oncol. 2003 Aug 15;21(16):3016-24. doi: 10.1200/JCO.2003.12.046. Epub 2003 Jul 1. PMID 12837811
- [Background] Tan EH, Rolski J, Grodzki T, Schneider CP, Gatzemeier U, Zatloukal P, Aitini E, Carteni G, Riska H, Tsai YH, Abratt R. Global Lung Oncology Branch trial 3 (GLOB3): final results of a randomised multinational phase III study alternating oral and i.v. vinorelbine plus cisplatin versus docetaxel plus cisplatin as first-line treatment of advanced non-small-cell lung cancer. Ann Oncol. 2009 Jul;20(7):1249-56. doi: 10.1093/annonc/mdn774. Epub 2009 Mar 10. PMID 19276396
- [Background] Yang JJ, Zhou Q, Liao RQ, Huang YS, Xu CR, Wang Z, Wang BC, Chen HJ, Wu YL. Nedaplatin/Gemcitabine Versus Carboplatin/Gemcitabine in Treatment of Advanced Non-small Cell Lung Cancer: A Randomized Clinical Trial. Chin J Cancer Res. 2012 Jun;24(2):97-102. doi: 10.1007/s11670-012-0097-8. PMID 23359648
- [Background] Teramoto K, Asada Y, Ozaki Y, Suzumura Y, Nakano Y, Sawai S, Tezuka N, Inoue S, Fujino S. A phase II study of docetaxel plus nedaplatin in patients with metastatic non-small-cell lung cancer. Cancer Chemother Pharmacol. 2012 Oct;70(4):531-7. doi: 10.1007/s00280-012-1941-8. Epub 2012 Aug 5. PMID 22864949
- [Background] Naito Y, Kubota K, Ohmatsu H, Goto K, Niho S, Yoh K, Ohe Y. Phase II study of nedaplatin and docetaxel in patients with advanced squamous cell carcinoma of the lung. Ann Oncol. 2011 Nov;22(11):2471-2475. doi: 10.1093/annonc/mdq781. Epub 2011 Mar 4. PMID 21378204
- [Background] Oshita F, Yamada K, Kato Y, Ikehara M, Noda K, Tanaka G, Nomura I, Suzuki R, Saito H. Phase I/II study of escalating doses of nedaplatin in combination with irinotecan for advanced non-small-cell lung cancer. Cancer Chemother Pharmacol. 2003 Jul;52(1):73-8. doi: 10.1007/s00280-003-0615-y. Epub 2003 May 16. PMID 12750839
- [Background] Shirai T, Hirose T, Noda M, Ando K, Ishida H, Hosaka T, Ozawa T, Okuda K, Ohnishi T, Ohmori T, Horichi N, Adachi M. Phase II study of the combination of gemcitabine and nedaplatin for advanced non-small-cell lung cancer. Lung Cancer. 2006 May;52(2):181-7. doi: 10.1016/j.lungcan.2006.01.004. Epub 2006 Mar 24. PMID 16563558
- [Background] Sznol M. Blockade of the B7-H1/PD-1 pathway as a basis for combination anticancer therapy. Cancer J. 2014 Jul-Aug;20(4):290-5. doi: 10.1097/PPO.0000000000000056. PMID 25098290
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Background] Patel SP, Kurzrock R. PD-L1 Expression as a Predictive Biomarker in Cancer Immunotherapy. Mol Cancer Ther. 2015 Apr;14(4):847-56. doi: 10.1158/1535-7163.MCT-14-0983. Epub 2015 Feb 18. PMID 25695955
- [Background] Wimberly H, Brown JR, Schalper K, Haack H, Silver MR, Nixon C, Bossuyt V, Pusztai L, Lannin DR, Rimm DL. PD-L1 Expression Correlates with Tumor-Infiltrating Lymphocytes and Response to Neoadjuvant Chemotherapy in Breast Cancer. Cancer Immunol Res. 2015 Apr;3(4):326-32. doi: 10.1158/2326-6066.CIR-14-0133. Epub 2014 Dec 19. PMID 25527356
- [Background] Koukourakis MI, Giatromanolaki A, Brekken RA, Sivridis E, Gatter KC, Harris AL, Sage EH. Enhanced expression of SPARC/osteonectin in the tumor-associated stroma of non-small cell lung cancer is correlated with markers of hypoxia/acidity and with poor prognosis of patients. Cancer Res. 2003 Sep 1;63(17):5376-80. PMID 14500371
- [Background] Kurtul N, Eroglu C, Unal D, Tasdemir EA, Orhan O, Zararsiz G, Baran M, Kaplan B, Kontas O. Prognostic value of SPARC expression in unresectable NSCLC treated with concurrent chemoradiotherapy. Asian Pac J Cancer Prev. 2014;15(20):8911-6. doi: 10.7314/apjcp.2014.15.20.8911. PMID 25374228
- [Background] Huang Y, Zhang J, Zhao YY, Jiang W, Xue C, Xu F, Zhao HY, Zhang Y, Zhao LP, Hu ZH, Yao ZW, Liu QY, Zhang L. SPARC expression and prognostic value in non-small cell lung cancer. Chin J Cancer. 2012 Nov;31(11):541-8. doi: 10.5732/cjc.012.10212. Epub 2012 Oct 10. PMID 23114088
- [Background] Kato T, Miyamoto M, Kato K, Cho Y, Itoh T, Morikawa T, Okushiba S, Kondo S, Ohbuchi T, Katoh H. Difference of caveolin-1 expression pattern in human lung neoplastic tissue. Atypical adenomatous hyperplasia, adenocarcinoma and squamous cell carcinoma. Cancer Lett. 2004 Oct 8;214(1):121-8. doi: 10.1016/j.canlet.2004.04.017. PMID 15331180
- [Background] Sunaga N, Miyajima K, Suzuki M, Sato M, White MA, Ramirez RD, Shay JW, Gazdar AF, Minna JD. Different roles for caveolin-1 in the development of non-small cell lung cancer versus small cell lung cancer. Cancer Res. 2004 Jun 15;64(12):4277-85. doi: 10.1158/0008-5472.CAN-03-3941. PMID 15205342
- [Background] Ho CC, Kuo SH, Huang PH, Huang HY, Yang CH, Yang PC. Caveolin-1 expression is significantly associated with drug resistance and poor prognosis in advanced non-small cell lung cancer patients treated with gemcitabine-based chemotherapy. Lung Cancer. 2008 Jan;59(1):105-10. doi: 10.1016/j.lungcan.2007.07.024. Epub 2007 Sep 11. PMID 17850918
- [Background] Chen D, Shen C, Du H, Zhou Y, Che G. Duplex value of caveolin-1 in non-small cell lung cancer: a meta analysis. Fam Cancer. 2014 Sep;13(3):449-57. doi: 10.1007/s10689-014-9707-6. PMID 24609521
- [Result] Pao W, Girard N. New driver mutations in non-small-cell lung cancer. Lancet Oncol. 2011 Feb;12(2):175-80. doi: 10.1016/S1470-2045(10)70087-5. PMID 21277552